CLINICAL TRIAL: NCT05657340
Title: Video Head Impulse Test and Seasickness Susceptibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, Yoni Gutkovich, Dr, Medical Corps, Israel Defense Force
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IDF-1873-2018
Record Dates: First submitted 2022-12-11; First posted 2022-12-20 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Sea Sickness
Keywords: motion sickness; video head impulse test; vestibular testing; seasickness susceptibility
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- seasickness susceptible (Experimental): 43 seasickness susceptible maritime crewmembers underwent video-head impulse test
  Interventions: Diagnostic Test: Video-head impulse testing
- seasickness non-susceptible (Other): 43 seasickness non-susceptible maritime crewmembers underwent video-head impulse test
  Interventions: Diagnostic Test: Video-head impulse testing

INTERVENTIONS:
Diagnostic Test: Video-head impulse testing — Video-head impulse testing is a recent diagnostic bed-side test for evaluation of semi-circular canal function.

SUMMARY:
This a case control study on seasickness susceptibility. 86 healthy maritime personal were divided to seasickness susceptible and non susceptible groups based on a seasickness questionnaire (Golding) and motion sickness score.

All subjects from both groups underwent video head impulse testing (vHIT). VHIT parameters - gain, asymmetry ect were compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 healthy military naval subjects
* At least six month of active sailing.

Exclusion Criteria:

* A history of hearing loss
* Ear pathology observed at otoscopic examination
* A neck injury precluding head movement.
* Abnormal otoneurological examination findings
* Subject's withdrawal of informed consent.
* Failure to complete the video head impulse test.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
vHIT gain | Immediate
  measurement of semicircular canal function
paired semi-circular canal asymmetry | Immediate
  (|1st canal gain-2nd canal gain|)/(1st canal gain+2nd canal gain)

SECONDARY OUTCOMES:
anterior semicircular canal gain o ipsilateral horizontal canal gain | Immediate
  anterior semicircular canal gain o ipsilateral horizontal canal gain

CONTACTS AND LOCATIONS:
Locations (1):
- Israeli Naval Medical Institute, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No
Information will be available upon reasonable request from corresponding author

REFERENCES:
- [Derived] Gutkovich YE, Jamison A, Lagami D, Fonar Y, Siag K, Tal D. Video head impulse test and seasickness susceptibility. Exp Brain Res. 2025 Apr 16;243(5):119. doi: 10.1007/s00221-025-07078-9. PMID 40237844